CLINICAL TRIAL: NCT01553734
Title: Does Azithromycin Cause QT Prolongation in Hospitalized Patients With Severe Community Acquired Pneumonia?
Status: Completed | Type: Observational
Sponsor: HaEmek Medical Center, Israel (Other)
Responsible Party: Sponsor
Other Study IDs: EMC-130-11
Record Dates: First submitted 2012-03-11; First posted 2012-03-14 (Estimated); Last update posted 2016-08-31 (Estimated); Status verified 2016-08

CONDITIONS: Pneumonia
Keywords: QT prolongation; Azithromycin; macrolide; pneumonia; ECG changes
MeSH Terms: conditions — Pneumonia; Long QT Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The macrolide group of antibiotics can cause QT prolongation, and endanger the patient with life threatening arrythmias. QT prolongation caused by Azythromycin, a relatively new macrolide, is extremely rare, and was not reported in clinical trials. Our hypothesis is that patients hospitalized with severe community acquired pneumonia, usually with multiple comorbid conditions will have a higher rate of QT prolongation, compared to the clinical trials published

DETAILED DESCRIPTION:
Patients hospitalized with community aquired pneumonia will have their corrected QT measured daily during antibiotic therapy. Concomittant medications and electrolyte abnormalities that cause prolonged QT will be recorded

ELIGIBILITY:
Inclusion Criteria:

* Severe community acquired pneumonia
* treated with azithromycin
* age over 18 years

Exclusion Criteria:

* Azithromycin initiated before hospitalization
* technically undecipherable ECG
* Permanent pacemaker

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients hospitalized with severe community aquired pneumonia treated with azithromycin
Sampling Method: Non-Probability Sample
Enrollment: 148 (Actual)
Dates: Start 2012-03; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Corrected QT segment of ECG | Daily, at estimated peak antibiotic level, during index hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Lee H Goldstein, MD, Principal Investigator — Haemek Medical Center, Afula, Israel
Locations (1):
- HaEmek Medical Center, Afula, Israel

IPD SHARING:
Plan to Share IPD: No